CLINICAL TRIAL: NCT03115281
Title: World-wide Registry to Assess the STENTYS Xposition S for Revascularization of Coronary Arteries In Routine cliNical Practice
Brief Title: Registry to Assess the STENTYS Xposition S for Revascularization of Coronary Arteries In Routine cliNical Practice
Acronym: WIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Stentys (Industry)
Responsible Party: Sponsor
Other Study IDs: ST2016-02
Record Dates: First submitted 2017-03-24; First posted 2017-04-14 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Coronary Self Expanding Stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PCI — PCI

SUMMARY:
WIN is a prospective, observational multinational post-marketing registry designed to evaluate the safety and effectiveness of the XPOSITION S STENT used in routine clinical practice.

DETAILED DESCRIPTION:
WIN is a prospective, observational multinational post-marketing registry designed to evaluate the safety and effectiveness of the XPOSITION S stent used in routine clinical practice. Subjects with coronary artery disease, including patients with chronic stable angina, silent ischemia and acute coronary syndrome, who qualify for elective percutaneous coronary interventions suitable for a self-expanding stent, can be included in the registry.

This registry will allow collecting data, and provide substantial information in a real world setting on patients with indications like lesions in vessels with diameter variance, large vessels, left main coronary artery, bifurcations, ectatic vessels, ...

WIN will enroll 750 patients from approximately 30 sites.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Presence of de novo coronary artery stenosis of ≥50% in a coronary artery suitable for implantation of the XPOSITION S STENT;
3. Vessel reference vessel diameter > 2.5 mm and ≤ 6.0 mm without excessive tortuosity or diffuse distal disease;
4. The target lesion is suitable for a drug-eluting self-expanding stent indication, as assessed by investigator;
5. The target lesion is 10mm or longer;
6. The patient has been fully informed of the study, written informed consent as approved by the applicable Ethics Committee.

Exclusion Criteria:

* Known pregnancy or breastfeeding; 2. Known contraindication or hypersensitivity to any stent components, any PCI-related material or drug.

  3. Concurrent medical condition with a life expectancy < 12 months; 4. Currently participating in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with this study endpoints; 5. Subjects undergoing cardiopulmonary resuscitation or in cardiogenic shock 6. Treatment of in-stent restenosis at target lesion; 7. Use of bioabsorbable/bioresorbable stents 8. Target lesion in left main coronary artery is excluded only if any of the following conditions is met:
  1. Ostial left main lesion;
  2. Presence of severe calcifications
  3. Vessel diameter is smaller than 3.0mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with coronary artery disease, including patients with chronic stable angina, silent ischemia and acute coronary syndrome, who qualify for Percutaneous Coronary Interventions suitable for a self-expanding drug eluting stent. Patient must be over legal age, and sign an authorization form for collection, transfer and processing of personal data.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
TLF at 1 Year follow-up | 1 year follow-up post-procedure
  Target Lesion Failure (TLF), defined as cardiac death, Myocardial Infarction (MI) attributable to the Target Vessel (TV), clinically driven Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
TLF at 2 Year | 2 year follow-up post-procedure
  Target Lesion Failure (TLF), defined as cardiac death, Myocardial Infarction (MI) attributable to the Target Vessel (TV), clinically driven Target Lesion
TVF at 1 Year | 1 year follow-up post-procedure
  Target Vessel Failure (TVF) defined as cardiac death, Myocardial Infarction (MI) attributable to the Target Vessel (TV), clinically indicated Target Vessel Revascularization (TVR),
Acute success rates | From Index procedure up to hospital discharge (48 hours post procedure)
  1. Device Success: Attainment of < 20% final in-stent residual stenosis of the target lesion with the XPOSITION S;
  2. Lesion Success: Attainment of < 20% final in-stent residual stenosis of the target lesion using any percutaneous method;
  3. Procedure Success: TIMI grade 3 and no in-hospital MACE
Stent thrombosis | 1-year and 2-year follow-up post procedure
  Stent thrombosis (definite/probable) - Academic Research Consortium (ARC) definition

CONTACTS AND LOCATIONS:
Locations (2):
- OLVG, Amsterdam, Netherlands
- Kantonsspital, Sankt Gallen, Switzerland